CLINICAL TRIAL: NCT06229795
Title: Effect of Green Tea on Obese Pediatrics With Prediabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sylvia Yousry Kamel Megaly, Teaching assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Green tea on obese pediatrics
Record Dates: First submitted 2024-01-09; First posted 2024-01-29 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: PreDiabetes
Keywords: Prediabetes, green tea, pediatrics, children, insulin resistance
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Metformin 500 mg tablet once daily and Green tea 300 mg film coated tablet three times daily.
  Interventions: Drug: Green Tea Leaf Extract Decaffeinated; Drug: Metformin Hydrochloride 500 MG
- Control (Active Comparator): Metformin 500 mg tablet once daily
  Interventions: Drug: Metformin Hydrochloride 500 MG

INTERVENTIONS:
Drug: Green Tea Leaf Extract Decaffeinated — 300 mg film coated tablet
  Arms: Intervention
Drug: Metformin Hydrochloride 500 MG — 500 mg tablet

SUMMARY:
The aim of this research is to evaluate the safety and efficacy of green tea in obese pediatrics with prediabetes versus the metformin therapy alone that is given to these patients. The primary outcome is to tackle the insulin resistance in these patients to prevent the deterioration of prediabetes to type 2 diabetes. The assessment of the effect on insulin resistance by using homeostatic model assessment for insulin resistance (HOMA-IR levels) as well as the effect on blood glucose levels and glycated hemoglobin. The other primary outcome is to observe the effect of the intervention on the lipid profile, leptin and adiponectin. The secondary outcome is to determine the effect of green tea on the oxidative and inflammatory markers and to evaluate its safety and efficacy. The study design is prospective parallel randomized open- label controlled interventional clinical trial that will be conducted in El-Demerdash hospital children's endocrinology unit. The patients who fit the inclusion criteria will be educated about the study protocol and will be required to sign a written informed consent. The inclusion criteria are: children whose age is between 10 to 18, whose HOMA-IR >2.5, BMI >= 95th percentile and have no sensitivity towards green tea and willing to sign informed consent. Patients who have causes of endogenous obesity will be excluded and those who have any other comorbid conditions. All patients fulfilling the inclusion criteria will be randomly assigned by simple randomization into either Group 1 (Control group): Consists of 45 patients who will receive their conventional therapy which is Metformin 500 mg film coated tablets (Glucophage).

Group 2 (Interventional group): Consists of 45 patients who will receive Green Tea 300 mg (Green tea 300 mg film coated tablets Mepaco Egypt) thrice daily + Metformin 500 mg film coated tablets (Glucophage). At baseline the following parameters will be collected during patients' interview and from patients' files: Demographic data as age, sex, weight and height (BMI), family history, medical history, medication history. The following laboratory' measurements will be tested at baseline and at the end of study (4 months): fasting plasma glucose, fasting plasma insulin, homeostatic model assessment for insulin resistance, homeostatic model assessment for β-cell function, lipid profile, leptin, adiponectin, malondialdehyde, liver functions, kidney functions, c-reactive protein, nuclear factor kappa beta.

Patients will be educated about the side effects and/or adverse effects of green tea, where safety and tolerability will be monitored by reporting the incidence of any side effect and /or adverse effect such as liver problems, yellowing of the color of skin or white of the eyes or stomach pain. Participants will be followed up during the study period every week through clinic visits and by phone in order to assure compliance as well as monitoring of incidence of any side/adverse effects and informing the patients who to handle it.

ELIGIBILITY:
Inclusion Criteria:

1. Homeostatic Model Assessment for Insulin Resistance (HOMA IR) >2.5
2. BMI >= 95th percentile according to CDC percentile charts
3. Age from 10 to 18 years.
4. Willing to sign a written informed consent through their caregivers.
5. Absence of sensitivity and/or known allergies for green tea.

Exclusion Criteria:

1. Homeostatic Model Assessment for Insulin Resistance (HOMA IR) <2.5
2. Endogenous obesity eg; thyroid dysfunction and adrenal glands dysfunction.
3. Presence of any other comorbidities as: cardiovascular, renal, liver etc…

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2023-11-12 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Effect on | At 0 weeks then after 16 weeks
  Homeostatic model assessment for insulin resistance (HOMA-IR)
Effect on | At 0 weeks then after 16 weeks
  Glycated hemoglobin (HbA1c)

SECONDARY OUTCOMES:
Effect on | At 0 weeks then after 16 weeks
  lipid profile
Effect on | At 0 weeks then after 16 weeks
  leptin
Effect on | At 0 weeks then after 16 weeks
  adiponectin
Effect on | At 0 weeks then after 16 weeks
  Malondialdehyde (MDA) oxidative stress marker
Effect on | At 0 weeks then after 16 weeks
  Nuclear factor kappa beta (NF-KB) inflammatory marker
Effect on | At 0 weeks then after 16 weeks
  Number of participants with treatment related adverse effects by using side effects card given to patients and performing liver function tests AST/ALT

CONTACTS AND LOCATIONS:
Locations (1):
- El-Demerdash hospital, Cairo, Egypt